CLINICAL TRIAL: NCT04447105
Title: Randomized Controlled Trial of the Effect of General Anesthetics on Postoperative Recovery After Minimally Invasive Nephrectomy (REGAIN Trial)
Brief Title: Comparison of Postoperative Recovery Between TIVA and Inhalation Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003-177-1113
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Enhanced Recovery After Surgery
Keywords: quality of recovery after surgery; anesthetic method
MeSH Terms: interventions — Propofol; Anesthesia, Inhalation; Desflurane

STUDY DESIGN:
Intervention Model Description: A prospective randomized single-blinded study
Who Masked: Participant
Masking Description: Patients will receive general anesthesia, therefore they can not know their anesthetic method.
  Physicians involved in this study will investigate the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Experimental): Patients receiving total intravenous anesthesia with propofol.
  Interventions: Drug: total intravenous anesthesia with propofol
- Desflurane group (Active Comparator): Patients receiving inhalation anesthesia with desflurane.
  Interventions: Drug: inhalation anesthesia with desflurane

INTERVENTIONS:
Drug: total intravenous anesthesia with propofol — In the TIVA group, general anesthesia is induced and maintained with a target-controlled infusion of propofol using infusion pump (Orchestra®; Fresenius Vial, Brezins, France). In both groups, remifentanil is continuously infused throughout the surgery for balanced anesthesia, adjusted to maintain arterial pressure.
  Other Names: TIVA group
  Arms: TIVA group
Drug: inhalation anesthesia with desflurane — In the desflurane group, anesthesia is induced with propofol 1-2 mg/kg and maintained with desflurane (5-7 vol %). In both groups, remifentanil is continuously infused throughout the surgery for balanced anesthesia, adjusted to maintain arterial pressure.
  Other Names: DES group
  Arms: Desflurane group

SUMMARY:
This prospective, randomized, single-blinded study is designed to compare the postoperative quality of recovery between propofol based total intravenous anesthesia and desflurane in patients undergoing minimally invasive nephrectomy. We hypothesize that propofol based total intravenous anesthesia can significantly improve the quality of recovery after surgery in patients with minimally invasive nephrectomy.

DETAILED DESCRIPTION:
Adult patients undergoing elective laparoscopic or robotic assisted nephrectomy are randomly allocated to receive propofol based total intravenous anesthesia (n=75) or desflurane (n=75). The quality of recover after surgery using the QoR-15K was assessed by a investigator at postoperative day (POD) 1, 2, and 3. The primary outcome is the QoR-15K at POD 1, 2, and 3 after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparoscopic or robotic assisted nephrectomy under general anesthesia
* American Society of Anesthesiologists (ASA) physical classification I-II
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Do not understand our study
* American Society of Anesthesiologists (ASA) physical classification III or more
* Allergies to anesthetic or analgesic medications
* Chronic pain, chronic analgesic or antidepressant or anticonvulsant use
* Medical or psychological disease that can affect the treatment response
* Patients who receive mechanical ventilation more than 2 hours after surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
quality of recovery | at 24 hours, 48 hours, 72 hours postoperatively
  Change in the QoR-15K score from 24 hours to 72 hours postoperatively

SECONDARY OUTCOMES:
Postoperative pain score | at 24 hours, 48 hours, 72 hours postoperatively
  Change in the pain severity measured by the 11-pointed numeric rating scale (0: none/10: worst pain) pain score at resting/movement from 24 hours to 72 hours postoperatively
Postoperative nausea and vomiting during the first 24 hours postoperatively | during the first 24 hours postoperatively
  Incidence of postoperative nausea and vomiting (%)
Postoperative nausea and vomiting during the 24-48 hours postoperatively | during the 24-48 hours postoperatively
  Incidence of postoperative nausea and vomiting (%)
Postoperative nausea and vomiting during the 48-72 hours postoperatively | during the 48-72 hours postoperatively
  Incidence of postoperative nausea and vomiting (%)
Total fentanyl consumption during the first 24 hours postoperatively | during the first 24 hours postoperatively
  Change in the postoperative fentanyl consumption (mcg) via IV patient controlled analgesia from 24 hours to 72 hours postoperatively
Total fentanyl consumption during the 24-48 hours postoperatively | during the 24-48 hours postoperatively
  Change in the postoperative fentanyl consumption (mcg) via IV patient controlled analgesia from 24 hours to 72 hours postoperatively
Total fentanyl consumption during the 48-72 hours postoperatively | during the 48-72 hours postoperatively
  Change in the postoperative fentanyl consumption (mcg) via IV patient controlled analgesia from 24 hours to 72 hours postoperatively
Quality of life at early post-discharge | day before surgery and at 3 weeks after discharge
  Change in the Quality of life measured using the EuroQoL 5-dimension 5-level scale (EQ-5D-5L) from baseline to early-postdischarge phase

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee WK, Kim MS, Kang SW, Kim S, Lee JR. Type of anaesthesia and patient quality of recovery: a randomized trial comparing propofol-remifentanil total i.v. anaesthesia with desflurane anaesthesia. Br J Anaesth. 2015 Apr;114(4):663-8. doi: 10.1093/bja/aeu405. Epub 2014 Dec 10. PMID 25500679